CLINICAL TRIAL: NCT02380339
Title: A Combined Biofeedback-virtual Reality System for Reduction of Fear of Hypoglycemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0098-14-HMO-CTIL
Record Dates: First submitted 2015-03-02; First posted 2015-03-05 (Estimated); Last update posted 2019-09-11 (Actual); Status verified 2019-08

CONDITIONS: Hypoglycemia; Type One Diabetes
MeSH Terms: conditions — Hypoglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psych-Educational and Bio Feedback (BF_ (Active Comparator): Participants in the control group will undergo Psych-Educational and BF sessions in which they will receive information about FOH and about ways of coping with FOH and BF training. More specifically, they will learn about factors associated with FOH, behavioral manifestations of FOH, negative consequences of these behavioral manifestations and about ways of coping with FOH. They will be instructed to practice BF for 15 minutes, at home for 5 initial training sessions during a week. After which they will receive another session of BF training and will be instructed to practice it at home for 10 sessions course, (5 weekly sessions for 2 weeks). Each session will be for 15 minutes.
  Interventions: Behavioral: Psych-Educational and BF sessions
- Psych-Educational session and virtual reality (VR) (Experimental): Participants in the intervention group will receive Psych-Educational session as the control group and in addition they will participate in training for VR system and will be asked to use it at home for 5 initial training sessions during a week. During this week, they will practice reducing their GSR levels as indicated by the BF device. Following this they will receive a combined biofeedback-virtual reality system and use it at home for a 10 sessions course, (5 weekly sessions for 2 weeks). Each session will be for 15 minutes.
  Interventions: Behavioral: Psych-Educational session and virtual reality

INTERVENTIONS:
Behavioral: Psych-Educational session and virtual reality — Psych-Educational session and virtual reality
  Arms: Psych-Educational session and virtual reality (VR)
Behavioral: Psych-Educational and BF sessions — Psych-Educational and BF sessions
  Arms: Psych-Educational and Bio Feedback (BF_

SUMMARY:
Uncontrolled diabetes is associated with increased risk for micro-vascular complication. Hypoglycemia is one of the major barriers in achieving good glucose control. Hypoglycemia is associated with a range of unpleasant symptoms including palpitations, tremor, hunger, sweating, confusion, difficulties in thinking as well as other idiosyncratic symptoms. Fear of hypoglycemia (FOH) refers to phobic avoidance reactions associated with hypoglycemia FOH may increase behavioral attempts to avoid hypoglycemia including decreased consumption of insulin and/or increased consumption of carbohydrates, resulting in poor glycemic control and an increased risk of diabetic complication. In this study, the investigators present a novel system, which simultaneously employs BioFeedback and Virtual Reality in order to cope with fear of hypoglycemia.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetic patient, male and females above the age of 18.
* Patients with significant fear of hypoglycemia as indicated in the HFS-W (equals or greater than 3 on at least one of the item on the HFS-W ).

Exclusion Criteria:

Patient with severe hypoglycemia event in the last 6 months will be excluded. Patient with mental illness will be excluded

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Reduction of fear of hypoglycemia in type 1 diabetic patients as measured by reduction of 2 point on the HFS-W). pre-treatment and after two months post completion of treatment. | two months

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel, Jerusalem, Israel